CLINICAL TRIAL: NCT01281709
Title: Primary Care Physician's Wishes and Influencing Factors Toward Provision of Integrated Health Care
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Tai-Yuan Chiu, President of Taiwan Association of Family Medicine, Taiwan Association of Family Medicine
Other Study IDs: 201011019RC
Record Dates: First submitted 2011-01-20; First posted 2011-01-24 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2011-01

CONDITIONS: Attitude of Health Personnel

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This questionnaire-based study was focused on understanding primary care physician's wish toward provision of integrated health care, associated knowledge and attitude, and analysis of influencing factors affecting their choices.

DETAILED DESCRIPTION:
The population is aging rapidly in Taiwan. It has been estimated that 15 years from now, the elderly population will comprise over 20% of the general population. Within an aging population, the prevalence of chronic illnesses can be expected to increase, and these patients with multiple chronic illnesses will likely need a larger allocation of available resources with the national health care system. In contrast to a highly-specialized medical environment, integrated health care, with its multitude of health and medical services including diagnosis, treatment, convalescence, rehabilitation, and health promotion, can provide a more efficient synergism between the necessary aspects of delivery, supply, management and organization. Literature has shown that multi-disciplinary, well-managed chronic illness management can increase the convenience of patient medical visits and also decrease medical costs. To provide patients with multiple chronic illnesses more suitable, efficient, and higher quality medical care, and to decrease redundant or ill-advised medications or procedures, as well as to encourage medical systems to further incorporate integrated services to advance the ideal of holistic care, the Bureau of National Health Insurance issued the a decree on September 15th, 2009, named "Integrated care model and medical system-based integration plan". This questionnaire-based study was focused on understanding primary care physician's wish toward provision of integrated health care, associated knowledge and attitude, and analysis of influencing factors affecting their choices.

ELIGIBILITY:
Inclusion Criteria:

* The primary care physicians, who practicing western medicine, with the doctor licenses approved by the Department of Health in Taiwan

Exclusion Criteria:

* The subjects who are unable to complete the survey independently

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The primary care physicians who serve in the excecutive centers of their community medical groups
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-03 (Estimated); Study Completion 2011-04 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Tai-Yuan Chiu, Master, Study Chair — National Taiwan University Hospital (NTUH)